CLINICAL TRIAL: NCT02071290
Title: Effect of Remote Ischemic Conditioning on Neutrophil Function and the Immune-Inflammatory and Coagulation Profiles in Trauma Patients With Hemorrhagic Shock
Brief Title: Effect of Remote Ischemic Conditioning on Trauma Patients With Hemorrhagic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SMH-RIC-01
Record Dates: First submitted 2014-02-18; First posted 2014-02-25 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Hemorrhagic Shock
Keywords: Hemorrhagic Shock; Remote Ischemic Conditioning
MeSH Terms: conditions — Shock, Hemorrhagic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Remote Ischemic Conditioning (Sham Comparator): Sham inflation of pneumatic tourniquet pressure cuff at 0 mmHg on the thigh for 5 minutes and release for 5 minutes (repeated for 4 cycles) applied to trauma patients on arrival to hospital
  Interventions: Device: Pneumatic tourniquet
- Remote Ischemic Conditioning (Experimental): Inflation of pneumatic tourniquet pressure cuff at 250mmHg on the thigh for 5 minutes and release for 5 minutes (repeated for 4 cycles) applied to trauma patients on arrival to hospital
  Interventions: Device: Pneumatic tourniquet

INTERVENTIONS:
Device: Pneumatic tourniquet — Four cycles of brief occlusion of bloodflow to the thigh (5 minutes) followed by reperfusion (5 minutes) using a pneumatic tourniquet
  Remote Ischemic Conditioning

SUMMARY:
The purpose of the study is to evaluate whether remote ischemic conditioning is a safe and effective intervention to prevent the development of inflammation and coagulopathy in trauma patients with hemorrhagic shock.

DETAILED DESCRIPTION:
Dysfunction of vital organs is one of the major reasons why trauma victims die after sustaining a major injury, even though the organs themselves may not have been directly injured. The inability to clot blood as a result of inflammation further contributes to complications in a majority of these patients. One intervention proposed to protect against impaired organ function is called "Remote Ischemic Conditioning", wherein application of intermittent occlusion and release of blood flow to the arm by sequentially inflating and deflating a blood pressure cuff can protect against the development of distant organ injury and inflammation following a severe traumatic event. In a pilot study, we will investigate the effects of remote ischemic conditioning in trauma patients with hemorrhagic shock, with a view to evaluate its effects on the immune system and coagulation profiles, both of which are known to be deranged in these patients. These studies will potentially benefit patients and will serve as a proof of principle for the use of remote ischemic conditioning in the trauma setting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16 years of age or estimated weight ≥50kgs if age is unknown;
* Victim of blunt or penetrating trauma
* Hemorrhagic shock defined as:
* One or more episodes of systolic blood pressure ≤90mmHg at any time prior to enrollment into the study;
* An identified source of blood loss (abdomen, chest, pelvis/retroperitoneum, extremities, external) or
* Blood products (RBC, Platelets, Plasma, etc.) has been ordered to the trauma room.
* Admitted to St. Michael's Hospital directly from the scene of injury within 3 hours of the injury
* Application and completion of Remote Ischemic Conditioning (RIC) within 4 hours of the injury

Exclusion Criteria:

* Pregnancy
* Non-hemorrhagic shock (i.e. tension pneumothorax, cardiac tamponade, spinal shock, etc.)
* Major burns > 20% total body surface area
* Fracture of both lower extremities (i.e. traumatic amputation, fractures)
* Absence of vital signs prior to admission, ongoing CPR, possibly dead on admission or not expected to survive beyond a few hours.
* Injury in both legs (traumatic amputation, fractures, etc.)
* Patients with a systolic blood pressure above 200mmHg
* Patients treated with anticoagulants, antiplatelet therapy (Warfarin, Aspirin), steroids or with a known bleeding disorder or known abnormality of blood flow to the limb (if known)
* Patients with osteoporosis or other bone disorders, peripheral nerve injury, abnormal nerve supply, peripheral neuropathy (if known) or preexisting traumatic injury to the limb.
* Morbid obesity (largest cuff size won't fit)
* If RIC is done clinically before research protocol begins.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ori D Rotstein, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Leung CH, Rizoli SB, Trypcic S, Rhind SG, Battista AP, Ailenberg M, Rotstein OD. Effect of remote ischemic conditioning on the immune-inflammatory profile in patients with traumatic hemorrhagic shock in a randomized controlled trial. Sci Rep. 2023 Apr 29;13(1):7025. doi: 10.1038/s41598-023-33681-3. PMID 37120600

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Started | 25 | 25
Completed | 21 | 18
Not Completed | 4 | 7
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 3 | 5
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (17) | 40 (17) | 39 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 16 | 14 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Neutrophil Oxidative Burst Activity
Description: Change in neutrophil oxidative burst activity (dihydrorhodamine, DHR) over 24 hours from admission. Measured by flow cytometry using whole blood samples.
Time Frame: 0 (Admission), 1, 3, and 24 hours after intervention
Measure: Median (Inter-Quartile Range); unit: Median Fluorescence Intensity
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Median Fluorescence Intensity
  Admission | 302 [222 to 383] | 302 [223 to 652]
  1 Hour | 298 [235 to 366] | 268 [194 to 536]
  3 Hour | 229 [166 to 311] | 202 [144 to 384]
  24 Hour | 337 [257 to 559] | 461 [256 to 580]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.56, Mixed Models Analysis

2. Primary Outcome: Neutrophil Oxidative Burst Activity (PMA Stimulated)
Description: Change in PMA stimulated neutrophil oxidative burst activity (dihydrorhodamine, DHR) over 24 hours. Measured by flow cytometry using whole blood samples.
Time Frame: 0 (Admission), 1, 3, and 24 hours after intervention
Measure: Median (Inter-Quartile Range); unit: Median Fluorescence Intensity
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Median Fluorescence Intensity
  Admission | 28812 [18030 to 52662] | 14772 [10827 to 35370]
  1 Hour | 27041 [15717 to 44051] | 13044 [5789 to 32778]
  3 Hour | 19027 [7871 to 37239] | 8753 [4579 to 24316]
  24 Hour | 4680 [2394 to 13554] | 2667 [1483 to 5595]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.287, Mixed Models Analysis

3. Primary Outcome: Neutrophil Adhesion Molecule Expression (CD11b)
Description: Change in neutrophil adhesion molecule (CD11b) expression over 24 hours from admission. Measured by flow cytometry using whole blood samples.
Time Frame: 0 (Admission), 1, 3, 24 hours after intervention
Measure: Median (Inter-Quartile Range); unit: Median Fluorescence Intensity
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Median Fluorescence Intensity
  Admission | 5492 [3533 to 8415] | 4341 [2552 to 7786]
  1 Hour | 5108 [3453 to 7993] | 5808 [3345 to 10511]
  3 Hour | 5889 [3253 to 8720] | 6362 [4136 to 7197]
  24 Hour | 9998 [6385 to 12919] | 6013 [3464 to 9852]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.597, Mixed Models Analysis

4. Primary Outcome: Neutrophil Adhesion Molecule Expression (CD62L)
Description: Change in neutrophil adhesion molecule (CD62L) expression over 24 hours from admission. Measured by flow cytometry using whole blood samples.
Time Frame: 0 (Admission), 1, 3, and 24 hours after intervention
Measure: Median (Inter-Quartile Range); unit: Median Fluorescence Intensity
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Median Fluorescence Intensity
  Admission | 5913 [4959 to 6879] | 5556 [4084 to 6807]
  1 Hour | 5404 [4352 to 6502] | 5452 [4743 to 7090]
  3 Hour | 4414 [3965 to 5770] | 4995 [4196 to 5603]
  24 Hour | 3742 [3228 to 4704] | 3569 [2629 to 4891]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.307, Mixed Models Analysis

5. Primary Outcome: Endothelial Injury (Heparan Sulfate)
Description: Change in plasma levels of endothelial injury marker Heparan Sulfate over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, and 24 hours after intervention
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
ng/mL
  Admission | 6.7 [3.4 to 8.4] | 6.0 [3.3 to 9.5]
  1 Hour | 3.3 [2.2 to 7.2] | 4.9 [2.5 to 10.2]
  3 Hour | 3.3 [1.9 to 7.1] | 3.6 [3.1 to 8.3]
  24 Hour | 3.0 [1.9 to 5.8] | 3.7 [2.9 to 6.5]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.646, Mixed Models Analysis

6. Primary Outcome: Endothelial Injury (Hyaluronan)
Description: Change in plasma levels of endothelial injury marker Hyaluronan over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 20 | 16
ng/mL
  Admission | 45.9 [24.4 to 78.1] | 36.6 [18.9 to 79.1]
  1 Hour | 35.6 [21.3 to 65.1] | 43.1 [17.6 to 65.3]
  3 Hour | 19.2 [13.9 to 52.6] | 26.5 [13.3 to 43.2]
  24 Hour | 54.9 [38.1 to 103.3] | 67.1 [34.2 to 130.9]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.757, Mixed Models Analysis

7. Primary Outcome: Endothelial Injury (Syndecan-1)
Description: Change in plasma levels of endothelial injury marker Syndecan-1 over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, and 24 hours after intervention
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
ng/mL
  Admission | 25.3 [16.6 to 67.8] | 27.2 [13.7 to 79.3]
  1 Hour | 35.0 [18.5 to 57.9] | 31.6 [16.3 to 109.7]
  3 Hour | 39.4 [15.3 to 64.4] | 48 [24.4 to 86.4]
  24 Hour | 24.3 [17.9 to 55.6] | 38.3 [23.4 to 67.0]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.075, Mixed Models Analysis

8. Primary Outcome: Plasma TNF-α
Description: Change in plasma levels of inflammatory mediator TNF-α over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, and 24 hours after intervention
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
pg/mL
  Admission | 2.15 [1.39 to 3.05] | 2.67 [1.65 to 3.25]
  1 Hour | 1.97 [1.51 to 2.68] | 2.34 [1.89 to 3.43]
  3 Hour | 1.95 [1.71 to 3.37] | 2.15 [1.72 to 3.06]
  24 Hour | 2.59 [2.07 to 3.52] | 2.72 [2.11 to 3.60]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.967, Mixed Models Analysis

9. Primary Outcome: Plasma IL-6
Description: Change in plasma levels of inflammatory mediator IL-6 over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
pg/mL
  Admission | 7.73 [3.77 to 60.09] | 8.04 [4.04 to 30.89]
  1 Hour | 11.95 [6.99 to 98.23] | 21.62 [5.33 to 51.99]
  3 Hour | 18.77 [11.82 to 90.98] | 23.30 [8.92 to 109.82]
  24 Hour | 65.72 [13.74 to 133.73] | 51.56 [25.63 to 137.76]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.637, Mixed Models Analysis

10. Primary Outcome: Plasma IL-8
Description: Change in plasma levels of inflammatory mediator IL-8 over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
pg/mL
  Admission | 7.1 [3.11 to 11.50] | 4.56 [2.78 to 7.46]
  1 Hour | 6.63 [2.95 to 36.42] | 5.81 [3.01 to 14.83]
  3 Hour | 9.85 [4.2 to 53.45] | 7.98 [2.82 to 34.05]
  24 Hour | 15.12 [5.50 to 26.65] | 9.53 [4.97 to 35.91]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.664, Mixed Models Analysis

11. Primary Outcome: Plasma IL-10
Description: Change in plasma levels of anti-inflammatory mediator IL-10 over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
pg/mL
  Admission | 1.93 [0.89 to 17.8] | 3.61 [1.10 to 8.03]
  1 Hour | 5.88 [2.22 to 43.42] | 8.58 [1.85 to 21.70]
  3 Hour | 5.56 [1.33 to 11.27] | 6.20 [1.24 to 17.06]
  24 Hour | 3.15 [0.84 to 6.86] | 2.11 [0.90 to 11.47]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.661, Mixed Models Analysis

12. Primary Outcome: ROTEM EXTEM CT
Description: Change in ROTEM parameter Clotting Time (CT) over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Seconds
  Admission | 71 [61 to 89] | 65 [60 to 69]
  1 Hour | 64 [59 to 73] | 62 [58 to 69]
  3 Hour | 68 [60 to 85] | 59 [56 to 71]
  24 Hour | 66 [55 to 72] | 71 [64 to 73]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.916, Mixed Models Analysis

13. Primary Outcome: ROTEM EXTEM CFT
Description: Change in ROTEM parameter Clot Formation Time (CFT) over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Seconds
  Admission | 90 [74 to 136] | 73 [55 to 85]
  1 Hour | 96 [79 to 135] | 108 [73 to 127]
  3 Hour | 125 [91 to 148] | 103 [82 to 129]
  24 Hour | 102 [76 to 115] | 91 [84 to 130]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.437, Mixed Models Analysis

14. Primary Outcome: ROTEM EXTEM A10
Description: Change in ROTEM parameter A10 over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
mm
  Admission | 54 [44 to 59] | 56 [53 to 64]
  1 Hour | 52 [44 to 56] | 48 [43 to 56]
  3 Hour | 46 [42 to 54] | 51 [43 to 54]
  24 Hour | 52 [48 to 59] | 54 [47 to 56]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.353, Mixed Models Analysis

15. Primary Outcome: ROTEM EXTEM Alpha Angle
Description: Change in ROTEM parameter Alpha Angle over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Degrees
  Admission | 72 [65 to 75] | 75 [73 to 79]
  1 Hour | 71 [64 to 74] | 71 [65 to 76]
  3 Hour | 68 [63 to 74] | 69 [65 to 74]
  24 Hour | 73 [70 to 76] | 72 [68 to 76]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.99, Mixed Models Analysis

16. Primary Outcome: ROTEM EXTEM ML
Description: Change in ROTEM parameter maximum lysis (ML) over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: Percent
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Percent
  Admission | 6 [3 to 11] | 6 [5 to 12]
  1 Hour | 5 [1 to 6] | 4 [3 to 7]
  3 Hour | 4 [1 to 6] | 4 [3 to 7]
  24 Hour | 8 [6 to 12] | 7 [4 to 11]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.085, Mixed Models Analysis

17. Primary Outcome: Plasma D-Dimer
Description: Change in plasma D-Dimer levels over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 20 | 18
ug/mL
  Admission | 0.96 [0.26 to 7.78] | 1.56 [0.57 to 10.12]
  1 Hour | 0.59 [0.30 to 3.63] | 1.50 [0.71 to 10.04]
  3 Hour | 0.85 [0.37 to 3.14] | 1.53 [0.66 to 10.91]
  24 Hour | 1.64 [0.52 to 4.27] | 1.70 [0.60 to 3.83]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.371, Mixed Models Analysis

18. Primary Outcome: Plasma Protein C
Description: Change in plasma Protein C levels over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: U/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 20 | 18
U/mL
  Admission | 0.65 [0.50 to 0.82] | 0.71 [0.66 to 0.81]
  1 Hour | 0.62 [0.50 to 0.95] | 0.70 [0.58 to 0.81]
  3 Hour | 0.70 [0.54 to 0.92] | 0.74 [0.69 to 0.88]
  24 Hour | 0.82 [0.71 to 1.00] | 0.75 [0.66 to 0.98]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.106, Mixed Models Analysis

19. Primary Outcome: Plasma Fibrinogen
Description: Change in plasma fibrinogen levels over 24 hours from Admission
Time Frame: 0 (Admission), 1, 3, 24 hours
Measure: Median (Inter-Quartile Range); unit: g/mL
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 20 | 18
g/mL
  Admission | 1.65 [1.29 to 2.54] | 2.44 [1.81 to 2.81]
  1 Hour | 2.09 [1.34 to 2.64] | 2.41 [1.54 to 2.70]
  3 Hour | 2.11 [1.65 to 2.68] | 2.35 [1.88 to 2.70]
  24 Hour | 3.91 [2.93 to 4.26] | 3.55 [3.04 to 4.26]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.829, Mixed Models Analysis

20. Secondary Outcome: Ventilator Free Days
Description: Secondary clinical outcomes
Time Frame: up to 28 days or discharge
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Days | 27 [24 to 28] | 26 [24 to 28]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.323, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: ICU Free Days
Description: Secondary clinical outcomes
Time Frame: up to 28 days or discharge
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Days | 27 [23 to 28] | 25 [18 to 27]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.287, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Hospital Free Days
Description: Secondary clinical outcomes
Time Frame: up to 28 days or discharge
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Days | 24 [11 to 26] | 16 [7 to 22]
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.151, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Nosocomial Infections
Description: Secondary clinical outcomes
Time Frame: up to 28 days or discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Participants | 5 | 6
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.510, Chi-squared

24. Secondary Outcome: 24 Hour Mortality
Description: Secondary clinical outcomes
Time Frame: up to 28 days or discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Participants | 1 | 0
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.348, Chi-squared

25. Secondary Outcome: 28 Day Mortality
Description: Secondary clinical outcomes
Time Frame: up to 28 days or discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
Number analyzed (Participants) | 21 | 18
Participants | 1 | 1
Statistical Analysis 1: Comparison: Sham Remote Ischemic Conditioning vs Remote Ischemic Conditioning; Test type: Superiority; p = 0.911, Chi-squared

ADVERSE EVENTS:
Time Frame: up to 28 days or discharge
Description: Chart review by research staff
Arm/Group | Sham Remote Ischemic Conditioning | Remote Ischemic Conditioning
All-Cause Mortality (participants affected / at risk) | 1/21 | 1/18
Serious Adverse Events (participants affected / at risk) | 6/21 | 9/18
Other Adverse Events (participants affected / at risk) | 0/21 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Remote Ischemic Conditioning (N=21) | Remote Ischemic Conditioning (N=18)
Nosocomial infection (Infections and infestations) | 5 (5) | 6 (6)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Thromboembolism (Vascular disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Prolonged EMS transport time, transfers, and clinical procedures contributed to delayed application and completion of RIC, resulting in several patients exceeding the 4-hour inclusion criteria and were therefore excluded due to protocol violation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No